CLINICAL TRIAL: NCT04816461
Title: Boosting the Impact of Seasonal Malaria Chemoprevention (SMC) Through Simultaneous Screening and Treatment of SMC-Children's Roommates in Burkina Faso
Brief Title: Boosting the Impact of SMC Through Simultaneous Screening and Treatment of Roommates
Acronym: SMC-RST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRSS006
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Malaria; Malaria Prophylaxis; Mass Testing and Treatment
Keywords: Chemoprevention; Roommate screening and treatment
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMC+ roommates screening with standard HRP2-RDT and treatment with DHAPPQ if positive (Experimental): SMC+ roommates screening with standard HRP2-RDT and treatment with DHAPPQ if positive
  Interventions: Drug: Amodiaquine Sulfadoxine-Pyrimethamin administration; Drug: Dihydroartemisinin-Piperaquine; Diagnostic Test: Standard HRP2-RDT
- SMC alone (Active Comparator): No roommates screening and treatment
  Interventions: Drug: Amodiaquine Sulfadoxine-Pyrimethamin administration

INTERVENTIONS:
Drug: Amodiaquine Sulfadoxine-Pyrimethamin administration — SMC treatment
Drug: Dihydroartemisinin-Piperaquine — Roommates treatment if they are positive to malaria
  Arms: SMC+ roommates screening with standard HRP2-RDT and treatment with DHAPPQ if positive
Diagnostic Test: Standard HRP2-RDT — Roommates screening with standard HRP2-RDT
  Arms: SMC+ roommates screening with standard HRP2-RDT and treatment with DHAPPQ if positive

SUMMARY:
Malaria represents a major public health concern in sub-Sahara Africa. Seasonal malaria chemoprevention (SMC) is one of the largest preventive measures. It consists to administer Amodiaquine+Sulfadoxine-Pyrimethamine to children aged 3-59 months on a monthly basis during the peak malaria transmission season. Despite its implementation, the burden of malaria is still very high in children under five years old in Burkina Faso. This raises questions about other hidden factors that can negatively affect the effectiveness of SMC intervention. Huge effort aiming at preventing human-vector contact were deployed such as the large-scale distribution of insecticide treated bed nets. Healthy humans are only infected via mosquitos if there are parasites reservoir around. Yet, there is no strategy aiming at protecting healthy humans from parasites reservoir. Under these circumstances, multiples humans sharing the same habitat could continually entertain the transmission cycle despite adequate existing measures. This would obviously jeopardize the expected impact of the SMC and the global effort to control the disease. In such context, we postulate that screening and treating malaria SMC-children's roommates could greatly improve the impact of SMC intervention and reduce malaria transmission in endemic settings.

The goal of our study is to improve the impact of SMC intervention in terms of reducing malaria morbidity and mortality in children under five years. Primary objectives include assessing whether SMC + children's roommates screening and treatment with Dihydro-artemisinin-piperaquine (DHAPPQ) is more effective than current routine implementation of SMC alone as well as the assessment of the tolerance and safety of AQSP and DHAPPQ. Secondary objectives include the assessment of the impact of the new strategy on the circulating parasite population in terms of selection of resistant strains and the assessment of determinants such as adherence and acceptability of the strategy.

Methodology: The study will be carried out in the Nanoro health district catchment area in Burkina Faso. This will be a randomized superiority trial. The unit of randomization will be the household and all eligible children from a household will be allocated to the same study group to avoid confusion. Households with 3 - 59 months old children will be assigned to either (i) control group (SMC alone) or (ii) intervention (SMC+ roommates screening with standard HRP2-RDT and treatment if positive) . The sample size will be 526 isolated households per arm, i.e. around 1,052 children under CPS coverage and 1,315 roommates expected. They will be followed-up for 24 months to fully cover two consecutive malaria transmission seasons and then two SMC cycles. Children will be actively followed-up during the malaria transmission seasons while in the dry seasons the followed-up will be passive.

DETAILED DESCRIPTION:
Malaria represents a major public health concern in sub-Sahara Africa. According to the World Health Organization (WHO) nearly half of the world's population is exposed to malaria infection causing 400 000 deaths yearly worldwide. In Burkina Faso like in most of sub-Sahara Africa countries, malaria remains endemic with peaks during raining seasons. To reduce the burden of the disease in the country, Burkina Faso has subscribed to the Roll Back Malaria initiative and adopted several malaria control measures including the use of artemisininin-based combination therapies as first line treatment since 2005, the intermittent preventive treatment for pregnant women, the wide-scale distribution of long-lasting insecticide treated net, and seasonal malaria chemoprevention (SMC) for children under five years old. However, despite the implementation of these multiple interventions, Burkina Faso is ranked among the top 10 countries carrying the highest malaria burden. For instance, in 2018, over 10 million clinical episodes and 4294 deaths were reported in the country.

In such context, new strategies to complement the existing ones or to improve their impact are urgently needed in order to reduce malaria transmission. The project we propose aims at improving the impact of Seasonal malaria chemoprevention (SMC) intervention to achieve best impact in malaria control and elimination. SMC is one of the largest and reliable malaria preventive measures recommended by WHO and is known to reduce malaria morbidity by 30 to 83%. It involves the administration of antimalarial drugs (Amodiaquine+Sulfadoxine-Pyrimethamine - AQSP) to children aged 3-59 months on a monthly basis during the high transmission season. In Burkina Faso, SMC is implemented nationally from July to October each year by the NMCP with the support of its technical and financial partners such as Global Fund, WHO, Malaria Consortium, PMI, UNICEF….). SMC was firstly implemented in 2014 in 6 of the 70 sanitary districts of the country. Few years later almost national wide coverage (except in Ouagadougou i.e. 60 over 70) was reached in 2018 and the intervention was adequately delivered by community health workers. Since the adoption of this strategy, data assessing the real-life impact of this intervention in the country are rare. In 2018, Druetz et al reported a protective effect of 62% highlighting the potential of this intervention for malaria control in Burkina Faso though this protective effect remains far below the highest threshold of 83% reduction of malaria incidence expected from SMC intervention. We anticipate that holding SMC campaigns in the context of the Covid-19 combined with the fact that some parts of the country are prone to insecurity may be challenging. However, it is important to stress that the year 2020 SMC campaign has been fully implemented in the study area without any disturbance related to the Covid and/or security issue. In addition, the study area, Nanoro is located at 85 km from Ouagadougou the capital city in the Central West Region of Burkina Faso where we have not experienced any particular security issues so far. With respect to research activities, the CRUN has no records of setbacks in fulfilling such activities due to security issues. All the research activities initiated before the insecurity onset have continued uninterrupted.

Furthermore, the burden of malaria in children under five years old suggests that the expected impact of this promising intervention is not achieved. Indeed, children under five years old represented the most affected population accounting for about 90% of malaria cases. RDT confirmed malaria cases in the country moved from 1 219 975 cases in 2016 to 1 487 954, and to 1 509 931, in 2017, and 2018 respectively. In view of the actual trend it becomes obvious that despite the implementation of this strategy, the burden of the disease and associated mortality is still very high in children under five years old in Burkina Faso, confirming that the expected impact from this intervention is not achieved. This raises questions about other hidden factors that can negatively affect the effectiveness of SMC intervention. At the same time, huge effort aiming at preventing human-vector contact were deployed such as the large-scale distribution of insecticide treated bed nets (LLIN). The latter are distributed on the basis of two individuals per unit. However, while most of the bedroom in rural setting in Burkina Faso are not adequate for the fixation of several LLIN, more than two individuals per room is commonly observed. In addition, the frequent mosquito bites before sleeping time and changing mosquito behavior becoming more aggressive before and after sleeping time is of concern. The latter could explain a persisting malaria transmission within a relatively close environment despite full coverage in LLIN.

Nevertheless, with regard to the infestation cycle, healthy humans are only infected via mosquitos if there are parasites reservoir (symptomatic and asymptomatic careers including sub-patent parasitaemia) around. Yet, there is no strategy aiming at protecting healthy humans from parasites reservoir. Under these circumstances, multiples humans sharing the same habitat (room, household) could continually entertain the transmission cycle despite adequate existing measures such as the use of LLIN. For instance, children under SMC coverage live closely with their family members e.g. mother, father, siblings and other relatives, who are not targeted by any specific interventions. According to the Nanoro health demographic surveillance system, an average of 3 inhabitants per household was observed. Published literature on sleeping behavior reported that children mostly sleep with their mother or with mother + sibling. Attempts to improve the impact of SMC intervention includes its extension to children under ten years old which showed promising results in Senegal. However, parents and elder siblings (over ten) not covered by the SMC (implemented either in under 5 or extended to under 10) sharing the same habitat could be parasites reservoir infecting continually the vulnerable group under SMC coverage. This is particularly important in a context of low coverage and compliance to ITN. Indeed, according to the household survey results in 2018 from the word malaria report, 54.5% of the population in Burkina Faso had access to ITN while only 44.1 had slept under ITN last night. This phenomenon of continual infestation of children from parents and elder siblings would obviously jeopardize the expected impact of the SMC intervention and the global effort to control the disease.

Finally, drug pressure, especially in wide scale community-based intervention such as SMC could lead to a selection of less sensitive mutant strains that could compromise the effectiveness of the intervention in a long-term period. Therefore, sustainability of any intervention relies on its selection pressure on parasite population which need to be closely monitored.

All these aspects underlie the idea of this project which stands on the assumption that screening and treating (if positive) malaria SMC-children's roommates could greatly improve the impact of SMC intervention and reduce malaria transmission in endemic settings.

The proposed project will respond to a major public health concern by providing evidence of the efficacy of a new strategy which should necessarily complement the existing ones to achieve best impact in malaria control and elimination.

A superiority of the intervention over the routine implementation of SMC alone is expected. By preventing malaria transmission within a relatively closed environment (shared rooms), the project is life-saving and is in line with global effort toward the achievement of SDG3 by horizon 2030. Therefore, the project will greatly contribute to the reduction of malaria burden in terms of reduction of its morbidity and mortality in Burkina Faso. In addition, the project will also contribute indirectly to the economic development by reducing the burden of malaria, which constitute huge threats to economic development in the country. Moreover, it will have a significant impact at the individual and community levels through, reduced attendance in education; reduced working days lost due to the disease; reduced individual, household, and community incomes because of the costs allocated to treatments.

By relying on existing strategy (SMC), if successful, the project could be scaled up easily at country and regional level especially for other Sahelian countries with similar malaria transmission profile and where SMC is implemented as well such as Mali, Niger, Mauritania, etc.

Furthermore, if successful, the project will strengthen the capacity of IRSS/CRUN by offering training opportunities to young researchers as one PhD and two M.Sc. degrees are expected by the end of this project. Finally, as a collaborative project, its implementation will strengthen the links between the IRSS/CRUN and collaborating partners namely the NMCP and the WWARN.

In view of all these aspects, it is obvious that at the end of this study, we will have not only collected data to answer the specific aims of the project, but will have also created a strong and sustainable research platform able to answer any relevant health research problem in the Greater Sahel in the future.

Type of research:

This will be a randomized superiority trial in which children will be followed-up for two years. The unit of randomization will be the household and all eligible children from a household will be allocated to the same study group to avoid confusion. The household will be defined as follow: one of several individuals living together within a shared habitat (house) and sharing basic needs, especially kitchen, and which recognizes the authority of a single person regardless of his/her gender. Households with 3 - 59 months old children with at least one under 35 months of age living within the Nanoro Health and Demographic Surveillance System (HDSS) catchment area will be assigned to either (i) control group (SMC alone) or (ii) intervention (SMC+ roommates screening with standard HRP2-RDT and treatment if positive).

Study population :

The study population will be children under SMC coverage i.e. aged 3-59 months and their roommates (individual of all years) living within the Nanoro HDSS catchment area. Children will be followed-up for 24 months to fully cover two consecutive malaria transmission seasons and then two SMC cycles. Children who leave the bracket covered by the CPS, i.e. whose age exceeds 59 months during the follow-up will subsequently be considered as roommates. Before the implementation of the year 1 first SMC round, a list of potential eligible households will be drawn from the HDSS database. Home visits will be performed to confirm the presence of the children and to assess willingness of the parents/guardians to participate in the study as well as willingness of all the roommates to be screened and treated. Households with absent children or children whose parents/guardians and roommates are not willing to participate, will be replaced by other eligible households from the list. Enrolment of study participants will be made in parallel with the SMC first round after confirmation of the administration of the first dose of the SMC treatment.

Sample size:

The aim is to demonstrate that SMC + roommates screening (through ultra-sensible RDT or classic RDT) and treatment arm is superior to the SMC alone arm in reducing the incidence of malaria after 1 year. The sample size is estimated for testing difference between two malaria incidence rates.

The estimation is performed under the assumption that the average number of malaria episode per child aged between 3-59 months per year since the implementation of Seasonal Malaria Chemoprevention (SMC) in Nanoro health district varied between 1.38 and 1.76 (Annual statistic yearly book, 2016, 2017 and 2018). Sample size of 236 in each arm will give at least 80% to detect 20% decrease in the incidence of malaria from a baseline incidence rate in SMC arm between 1.5- 2.0 malaria cases per year, assuming one-sided test with significance level of 0.025.

To account for 10% study, drop-out rate for any reason, the sample size will increase to 263 in each arm.

Therefore, the final estimated sample size for this study is 526 households (with at least one child aged between 3-59 months). Assuming that each household will have an average of 2 children under SMC coverage, about 1052 children under SMC coverage are expected. The expected number of roommates is estimated at about 1315 (263x5) under the assumption that each household from the 2 interventions arms will have an average of 5 roommates.

Data will be analyzed with R software using the appropriate tests depending on the variables. Adherence of treatment and acceptability of the strategy (focus group discussion) will be assessed qualitatively.

ELIGIBILITY:
Inclusion Criteria:

* Single household (not sharing the same concession with other households) with children under SMC coverage (aged 3-59 months) with at least one child under 35 months of age,
* Household members residing within the HDSS catchment area,
* Willingness of roommates to be screened and treated,
* Ability to complete the study follow-up period,
* Written consent obtained from parents/guardian
* Written consent/assent obtained from roommates

Exclusion Criteria:

* Household with children under SMC coverage who did not receive the SMC (Amodiaquine-Sulfadoxine-Pyrimethamine) or sharing the same concession with other households
* Household with children under SMC coverage but at least one of his/her roommates refuse to be screened and treated (these children will still receive the SMC treatment as part of their routine malaria prevention policy)
* Severely ill individual at the time of enrolment including severe malaria,
* Known allergy to AQSP for children and DHAPPQ for roommates
* Planned travel or inability to complete the study follow-up,
* Participation to malaria vaccine trial
* Unwillingness to participate to the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The incidence of uncomplicated malaria in each intervention arm versus SMC alone arm | 1 year
  Incidence of uncomplicated malaria in each intervention arm versus SMC alone arm
The incidence of severe malaria in each intervention arm versus SMC alone arm | 1 year
  Incidence of severe malaria in each intervention arm versus SMC alone arm

SECONDARY OUTCOMES:
The incidence of adverse events in each intervention arm versus SMC alone arm | 5 months
  Incidence of adverse events in each arm

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherche en Sciences de la Santé/ Clinical Research Unit of Nanoro, Nanoro, Boulkiemdé, Burkina Faso

IPD SHARING:
Plan to Share IPD: Undecided